CLINICAL TRIAL: NCT04422522
Title: Prevalence of Fibromyalgia in the Rheumatology Outpatient Clinics in the UAE During the COVID-19 Pandemic: a Cross-sectional Study
Brief Title: Fibromyalgia During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abogamal, Professor, Al-Azhar University
Other Study IDs: AAGH-01
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Fibromyalgia, Primary
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
On 12 January 2020, the World Health Organization (WHO) confirmed that a novel coronavirus was the cause of a respiratory illness in a cluster of people in Wuhan City, Hubei Province, China, which was reported to the WHO on 31 December 2019.

There is evidence of a high prevalence of psychiatric comorbidities in Fibromyalgia (FM )(especially depression, anxiety, post-traumatic stress disorder), which are associated with a worse clinical profile.

In these challenging times of COVID-19, anxiety increased among the general population. Fibromyalgia patients are more at risk of developing anxiety in these difficult times. This might result in more frequent visits to the rheumatology clinics with an exacerbation of their chronic pain syndrome.

DETAILED DESCRIPTION:
The first confirmed case relating to the COVID-19 pandemic in the United Arab Emirates was announced on 29 January 2020.

On March 11, the World Health Organization (WHO) declared the global outbreak a pandemic. Many measures have been taken by the UAE government since the COVID-19 outbreak started hitting the region. From Mid March, the UAE had advised all citizens to restrict themselves to essential travel only and had implemented a curfew between 8 pm and 6 am every day starting from the end of March. On April 5th, UAE imposed a two-week lockdown to contain the COVID-19 pandemic and announced there will be disinfection drives.

Many awareness campaigns were initiated by rheumatologists through different media channels advising patients with rheumatic diseases to avoid clinics and hospitals unless they have an emergency. Some healthcare facilities started telemedicine services including rheumatology outpatient clinics. However, most of the clinics and hospitals have maintained open rheumatology clinics aiming to manage emergency cases.

Fibromyalgia (FM) is a chronic disorder characterized by widespread and chronic musculoskeletal pain and other frequent syndromes such as chronic fatigue sleep disturbance, cognitive impairment, irritable bowel disease, depression, and anxiety.

There is evidence of a high prevalence of psychiatric comorbidities in FM (especially depression, anxiety, post-traumatic stress disorder), which are associated with a worse clinical profile.

In these challenging times of COVID-19, anxiety increased among the general population. Fibromyalgia patients are more at risk of developing anxiety in these difficult times. This might result in more frequent visits to the rheumatology clinics with an exacerbation of their chronic pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 year
* Diagnosis of primary fibromyalgia
* Newly diagnosed and follow up patients are included
* Patients who have physically attended the rheumatology clinic during the study period.

Exclusion Criteria:

* Patients aged < 18-year-old
* Patients with inflammatory arthritis and associated FM (Secondary FM)
* Patients who didn't physically attend the rheumatology clinics (Those who used Phone calls and other telemedicine platforms).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the rheumatology outpatients clinics (OPD) during the COVID-19 lockdown period (2020)
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of FM patients | two months
  Number of FM patients in the rheumatology outpatient clinics during the COVID-19 lockdown period (2020)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abogamal, Principal Investigator — Al-Azhar Faculty of medicine- Cairo
Locations (1):
- Al-Azhar Faculty of medicine, Rheumatology Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided